CLINICAL TRIAL: NCT04608266
Title: A Multicenter Randomized Trial to Evaluate the Efficacy and Safety of Camostat Mesylate for the Treatment of SARS-CoV-2 Infection - COVID-19 in Ambulatory Adult Patients (CAMOVID)
Brief Title: CAMOVID : Evaluation of Efficacy and Safety of Camostat Mesylate for the Treatment of SARS-CoV-2 Infection - COVID-19 in Ambulatory Adult Patients
Acronym: CAMOVID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Scientific committee decision due SARS-CoV2 pandemic evolution with a decrease in inclusions and widespread distribution of vaccines
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200702
Record Dates: First submitted 2020-10-28; First posted 2020-10-29 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — camostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camostat mesylate (Experimental): Camostat mesylate, oral administration 600mg/day
  Interventions: Drug: Camostat Mesylate
- Placebo (Placebo Comparator): Placebo tablets, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Camostat Mesylate — Camostat mesylate, oral administration 600mg/day (2 x 100mg tablets every 8 hours) for 14 days
  Arms: Camostat mesylate
Drug: Placebo — Placebo tablets, oral administration 2 tablets every 8 hours for 14 days
  Arms: Placebo

SUMMARY:
The overall objective of the study is to determine the therapeutic effect and tolerance of Camostat mesylate, compared to placebo in adult patients with ambulatory COVID-19 disease, presenting with risk factors of severe COVID-19. Camostat mesylate is a serine protease TMPRSS2 (Transmembrane Serine Protease 2) inhibitor which has been successfully and safely used to treat pancreatitis-associated pain and post-operative reflux oesophagitis in Japan. More recently, it has been shown to inhibit SARS-CoV-2 viral entry and reduce infection of human primary pneumocytes and lung cell lines.

Camostat mesylate or placebo will be administered to consenting adult patients with virologically confirmed COVID-19, not requiring initial hospitalization. All patients will receive standard of care along with randomized treatments. Outcomes of included patients will be compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients with an increased risk of severe COVID-19 belonging to one or more of the following groups :

  * Age ≥ 50 years
  * Body Mass Index ≥ 30 kg/m²
  * Diabetes
  * Hypertension
  * Chronic renal failure (eGFR <60 mL/min)
  * Chronic heart disease
  * Asthma/Chronic Obstructive Pumonary Disease/Cystic fibrosis
  * Chronic liver disease
  * Chronic neurological disease
  * Solid organ transplant
  * Bone marrow transplant
  * Sickle cell anemia/ Major thalassemias
  * Active or currently treated or <1 year diagnosed cancer
  * Active or currently treated or <1 year diagnosed malignant blood disease
  * Immunosuppressive treatment observed for more than 1 month
* Laboratory confirmed SARS-CoV2 infection with mild COVID-19, fulfilling all the following criteria:

  * Positive SARS-CoV-2 RT-PCR nasal swab samples AND
  * Clinical symptoms and signs consistent with SARS-CoV2 infection including but not limited to, fever, upper respiratory tract infection signs, digestive signs, muscle pain, anosmia, dysgueusia…(1)
* Informed consent to participate to the trial
* Patients must be able and willing to comply with study visits and procedures

Exclusion Criteria:

* Initial need for hospitalization for COVID-19 management
* Pregnancy and breastfeeding
* Participation to another interventional drug trial
* Subject protected by law under guardianship or curatorship
* Absence of health insurance
* Known hypersensitivity to camostat mesylate
* Known person sharing the same household already included in the study
* Participation to another COVID-19 ambulatory interventional study
* Patients having completed a full SARS-CoV2 vaccine immunization procedure less than 4 weeks prior to COVID-19 diagnosis (last vaccine injection performed less than 4 weeks prior to COVID-19 diagnosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Hospitalization for COVID-19 deterioration or death without hospitalization | Day 21
  Proportion of patients hospitalized for COVID-19 deterioration or who died without hospitalization

SECONDARY OUTCOMES:
Adverse events | Day 21
  Number of patients with at least one adverse event
Serious adverse events | Day 21
  Number of patients with at least one serious adverse event
Investigational medication discontinuation | Day 21
  Number of patients who discontinued the investigational medication
Hospitalization for COVID-19 deterioration or death without hospitalization, evaluated by independent adjudication comittee | Day 21
  Proportion of patients hospitalized for COVID-19 deterioration (reviewed by independent adjudication comitter) or who died without hospitalization
Clinical improvement using the Word Health Organization (WHO) COVID-19 scale | Day 7, 14, 21
  WHO clinical scale: Uninfected - No clinical or virological evidence of infection: 0; Ambulatory - No limitation of activities: 1; Ambulatory - limitation of activities: 2; Hospitalized - no oxygen therapy: 3; Hospitalized - oxygen by mask or nasal prongs: 4; Hospitalized; oxygen by non invasive ventilation or High flow: 5; Intubation and Mechanical ventilation: 6; Mechanical ventilation + additional organ support (pressors, Renal replacement therapy, ECMO):7; Dead: 8
Need for intensive care | Day 21
  Proportion of patients admitted to an intensive care unit
Duration of hospitalization | Day 21
  Number of days alive without hospitalization up to day 21
Need for invasive mechanical ventilation for severe COVID-19 | Day 21
  Proportion of patients with initiation of invasive mechanical ventilation
Need for oxygen therapy for COVID-19 | Day 21
  Proportion of patients with initiation of oxygen therapy
Overall survival | Day 90
  Proportion of patients alive at day 90
Duration of symptoms | Day 21
  Number of days alive without symptoms at day 21
SARS-CoV-2 virological assessment | Day 7, 14, 21
  By Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) on nasal swab and droplet quantification of SARS-CoV2 ribonucleic acid-emia (RNAemia)
SARS-CoV-2 serological assessment | Day 7, 14, 21 and 90
  SARS-CoV2 antibodies quantification in blood
Peripheral blood lymphocyte phenotyping | Day 1, 14, 90
  Peripheral blood lymphocyte phenotyping with telomere length measurement
Acute kidney failure | Day 21
  Acute kidney failure defined as at least serum creatinine increase of 0.3mg/dl or 1.5-1.9 times baseline and/or oliguria < 0.5ml/kg/h
Renal function | Day 7, 14 and 21
  estimated glomerular filtration rate
Concentration of urea in blood | Day 7, 14 and 21
  Uricemia in mmol/L or mg/dL
Concentration of potassium in blood | Day 7, 14 and 21
  Kaliemia in mmol/L
Liver function | Day 7, 14 and 21
  Liver transaminases dosage on blood sample
Liver function (2) | Day 7, 14 and 21
  Gamma-glutamyl transferase (gamma-GT) dosage on blood sample

OTHER OUTCOMES:
Biobanking for biomarker assessment | Day 1, 7, 14, 21, 90
  Biobanking of blood samples for predictive biomarker assessment

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - AP-HP Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Sud Ile de France - Melun, Melun
  - AP-HP Hôpital Bichat, Paris
  - APHP - Saint Louis, Paris
  - Centre de Santé Richerand, Paris

IPD SHARING:
Plan to Share IPD: Undecided